CLINICAL TRIAL: NCT06878924
Title: Safety and Efficacy of Pulmonary Vein Isolation Using Pulsed-field Ablation (PFA) Combined with Either PFA-based Left Atrial Posterior Wall Isolation or Vein of Marshall Ethanol Ablation in Patients with Persistent Atrial Fibrillation
Acronym: SAVIOR
Status: Not yet recruiting | Type: Observational
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Other Study IDs: TCAI_SAVIOR
Record Dates: First submitted 2025-03-05; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Persistent AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Persistent AF patients receiving PVI (PFA)+ VoM alcohol ablation: PVI:
  General periprocedural guidance includes target activated clotting time (ACT) ≥350, catheter exchange ≤2, >10s spacing of consecutive applications, and minimization of number of PF applications per the recommended procedures below:
  For each pulmonary vein, a concentric ring of applications will be created using 12 (6 ostial and 6 antral) applications In case of visual gaps, additional 8 applications will be added
  PWI:
  Concentric overlapping ablations will be placed throughout the posterior wall deliberately. The catheter will be rotated once between a pair of applications; briefly, rotation is performed such that, post-rotation, the splines are situated midway between the splines' pre- rotation positions. The number of applications will be at the operator's discretion.
  VoM:
  VoM alcohol ablation procedure will be conducted before the catheter ablation. VoM will be visualized by coronary sinus venography, cannulated with an angioplasty wire and balloon and 1 cc of 98% ethanol will
- PFA-based PVI+ left atrial posterior wall isolation: PVI:
  General periprocedural guidance includes target activated clotting time (ACT) ≥350, catheter exchange ≤2, >10s spacing of consecutive applications, and minimization of number of PF applications per the recommended procedures below:
  For each pulmonary vein, a concentric ring of applications will be created using 12 (6 ostial and 6 antral) applications In case of visual gaps, additional 8 applications will be added
  PWI:
  Concentric overlapping ablations will be placed throughout the posterior wall deliberately. The catheter will be rotated once between a pair of applications; briefly, rotation is performed such that, post-rotation, the splines are situated midway between the splines' pre- rotation positions. The number of applications will be at the operator's discretion.

SUMMARY:
This study is designed to directly compare the safety and efficacy of PFA-based PVI+PWI vs PFA-based PVI+ VoM alcohol ablation in patients with Persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent AF; 1st or redo ablation with PVI-only in the earlier procedure
* Willing to provide informed consent
* Age: 18-85 years

Exclusion Criteria:

* • Previous PWI or VoM ablation procedure

  * Left ventricular ejection fraction <40%
  * Left atrial thrombus
  * Myocardial infarction within last 60 days
  * Cardiac surgery in the last 6 months
  * Advanced renal failure
  * Life expectancy <1 year
  * Pregnant women
  * Unable or unwilling to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persistent atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia: any episode of AF/AT longer than 30 sec off-AAD, after the 2-month blanking period | 1 year

SECONDARY OUTCOMES:
• Arrhythmia-free on previously ineffective AAD without any dose-escalation | 1 year

IPD SHARING:
Plan to Share IPD: Yes
In order to protect the privacy of the patients, only analyzed data will be shared for research purpose, at the discretion of the PI